CLINICAL TRIAL: NCT02692131
Title: Comparison of Two Different Methods of Obtaining Strain by Perioperative Transesophageal in Patients Undergoing Coronary Artery Bypass Grafting : An Observational Study
Brief Title: Comparison of Two Methods of Strain by Perioperative Transesophageal Echo in CABG : An Observational Study
Acronym: Strain
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Alok Kumar, Fellow, Cardiac Anaesthesia, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK/2496/study
Record Dates: First submitted 2016-02-16; First posted 2016-02-25 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Artery Disease
Keywords: Left Ventricle strain, speckle strain
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Speckle strain: All adult patients undergoing on pump CABG Surgery.
- Tissue doppler strain: All adult patients undergoing on pump CABG Surgery

SUMMARY:
There is an increasing need for diagnostic modalities able to objectively quantify myocardial function. Quantification of regional myocardial function with ultrasound is challenging on its own. Visual assessment of wall motion and thickening requires extensive training [1] and remains highly subjective [2]. Tissue deformation imaging is a recently introduced technique which enables the objective assessment of regional myocardial deformation assessed by ultrasound based strain and strain rate using Doppler Tissue Imaging or Speckle tracking. There are limited number of studies comparing the myocardial deformation parameters (i.e. Strain and Strain rate) by 2 different echocardiographic techniques viz Doppler tissue imaging and Speckle tracking in the perioperative period. In this study, we plan to study the above said parameters in patients undergoing coronary artery bypass grafting using transesophageal echocardiography and correlate these parameters with cardiac output by thermodilution method using pulmonary artery catheter.

DETAILED DESCRIPTION:
The study will be conducted in the Department of Anaesthesiology and Intensive Care, Advanced Cardiac Centre, Post Graduate Institute Medical Education Research, Chandigarh after obtaining institutional ethical committee clearance. Fifty patients scheduled for coronary artery bypass grafting (CABG) will be included in the study. An informed written consent will be taken from all the patients.

Anaesthesia technique All patients will be examined a day prior to surgery. Baseline data including preoperative physical status, haemogram, biochemistry, preoperative transthoracic echocardiography and coronary angiography data will be noted. A standard anaesthesia technique will be used for all the patients. Inside the operating room, electrocardiography (ECG), pulse oximetry and noninvasive blood pressure (NIBP) will be applied. Anaesthesia will be induced with fentanyl 5 - 10 µg/kg/ body weight and propofol titrated to loss of response to verbal commands followed by endotracheal intubation facilitated by vecuronium 0.1mg/kg. A 20 gauge arterial catheter will be inserted in left radial artery and right internal jugular vein will be cannulated with triple lumen catheter for central venous access and pulmonary artery catheter for haemodynamic assessment. A baseline transthoracic echocardiogram will be performed after induction of general anaesthesia. After induction of general anaesthesia , a TEE probe (GE Medical Systems, Horten, Norway) will be introduced. Anaesthesia will be maintained by isoflurane, intravenous morphine (intermittent boluses; total 0.5 mg/kg during surgery) and vecuronium boluses. All patients will undergo CABG under cardiopulmonary bypass (CPB) support. Total cardiopulmonary bypass time and Aortic cross clamp time will be noted. Patients will be shifted to cardiac surgical intensive care unit (ICU) and electively ventilated. Decision on extubation and inotrope support will be left to attending intensivist.

Echocardiography data After induction of general anaesthesia, a comprehensive transesophageal echocardiogram will be performed using probe of the GE vivid E9 echocardiography system (GE Medical Systems, Hortein, Norway) in all the patients.

The following parameters will be noted before instituting CPB and after weaning from CPB and achievement of stable haemodynamics:

1. 2 dimensional Left ventricular ejection fraction using Simpson's method from midesophageal 4 chamber and midesophageal 2 chamber views.
2. 3 dimensional Left ventricular ejection fraction from midesophageal 4 chamber and midesophageal 2 chamber views.
3. Doppler tissue imaging derived regional and global longitudinal strain from midesophageal 4 chamber, midesophageal 2 chamber and midesophageal long axis views.
4. Speckle track imaging derived regional and global longitudinal strain from midesophageal 4 chamber, midesophageal 2 chamber and midesophageal long axis views.

An average of 3 readings over 3 different cardiac cycles will be used for above parameters.

ELIGIBILITY:
Inclusion Criteria:

* > 18 yrs
* On pump CABG

Exclusion Criteria:

* < 18 yrs
* other on pump cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (> 18 yrs) patients undergoing on pump CABG.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Correlation between left ventricle strain measured by Doppler tissue imaging and speckle tracking using transesophageal echocardiography in patients undergoing coronary artery bypass surgery. | Intraoperatively before going on bypass and 30 mins after coming off bypass.

CONTACTS AND LOCATIONS:
Overall Officials: Banashree mandal, MD, DM, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided